CLINICAL TRIAL: NCT04778800
Title: A Dose Exploration Study of Almonertinib for Epidermal Growth Factor Receptor(EGFR)-Mutant Non-small-cell Lung Cancer(NSCLC) Patients With Newly Diagnosed or Recurrent Brain/Leptomeningeal Metastasis (ARTISTRY)
Brief Title: A Dose Exploration Study of Almonertinib for EGFRm NSCLC Patients With Brain/Leptomeningeal Metastasis (ARTISTRY)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, wanghj, associate chief physician, Henan Cancer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-HS-006
Record Dates: First submitted 2021-01-27; First posted 2021-03-03 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: NSCLC; Brain Metastases; Leptomeningeal Metastasis
MeSH Terms: conditions — Brain Neoplasms; Meningeal Carcinomatosis | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- almonertinib 110mg PO once daily (Experimental)
  Interventions: Drug: almonertinib
- almonertinib 160mg PO once daily (Experimental)
  Interventions: Drug: LM-first line treatment
- almonertinib 220mg PO once daily (Experimental)
  Interventions: Drug: LM-second line treatment

INTERVENTIONS:
Drug: almonertinib — Patients was given a standard dose of 110mg/day of almonertinib, orally, and the first efficacy evaluation was carried out 4 weeks later. If the patient's lungs and/or other parts of the disease (PD) progress, then leave the group to receive other treatment; if the patient's lungs If the brain and other parts are stable or relieved and the brain has not progressed, continue the original dose treatment, and evaluate the effect every 8 weeks. Until the patient's lungs and/or other parts progress (PD), then leave the group to receive other treatment; if If the patient's lungs and other parts are stable or relieved and the brain is progressing, the dose of almonertinib can be increased to 165mg/day, orally ± radiotherapy (the investigator's decision), and then the efficacy will be evaluated every 8 weeks until the patient's lungs and/ Or there is progress (PD) in other parts, then the group will receive other treatment.
  Arms: almonertinib 110mg PO once daily
Drug: LM-first line treatment — Patients were given a standard dose of almonertinib 110 mg/day, orally, and the first efficacy evaluation was performed 4 weeks later. If there was no disease progression in two consecutive evaluations, the dose of almonertinib was increased to 165 mg /Day, oral ± radiotherapy (decided by the investigator), continue to evaluate the efficacy every 4 weeks until the patient progresses; if there is no disease progression in two consecutive assessments, the dose of almonertinib is increased to 220 mg/day, orally ± Radiotherapy treatment (determined by the investigator), continue to evaluate the efficacy every 4 weeks until the patient progresses.
  Arms: almonertinib 160mg PO once daily
Drug: LM-second line treatment — Patients were given a standard dose of almonertinib 110 mg/day, orally, and the first efficacy evaluation was performed 4 weeks later. If there was no disease progression in two consecutive evaluations, the dose of almonertinib was increased to 165 mg /Day, oral ± radiotherapy (decided by the investigator), continue to evaluate the efficacy every 4 weeks until the patient progresses; if there is no disease progression in two consecutive assessments, the dose of almonertinib is increased to 220 mg/day, orally ± Radiotherapy treatment (determined by the investigator), continue to evaluate the efficacy every 4 weeks until the patient progresses.
  Arms: almonertinib 220mg PO once daily

SUMMARY:
Almonertinib is a three-generation epidermal growth factor receptor tyrosine kinase inhibitor(EGFR-TKI), which has shown competitive potential in the second-line treatment against first-generation TKIs. This study aims to explore the efficacy and safety of different doses of almonertinib in the first-line and second-line treatment of brain metastases/meningeal metastases in NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

Queue 1

1. Male or female,age at least 18 years ;
2. Histologically confirmed patients with NSCLC brain metastases (including patients who have relapsed after previous treatment or newly diagnosed);
3. There must be at least one measurable brain lesion that has not been locally treated at the time of enrollment;
4. Patients who have not received other systemic treatment after the diagnosis of NSCLC brain metastasis, or patients who have received neoadjuvant therapy, adjuvant therapy, concurrent radiotherapy and chemotherapy, and local radiotherapy for more than 6 months;
5. Tumor tissue samples or blood are confirmed to be EGFR sensitive mutations (including exon 19 deletion or L858R) by ARMS;
6. The Eastern Cooperative Oncology Group (ECOG) physical status score is 0-2 and has not deteriorated in the previous 2 weeks, with a minimum expected survival of 12 weeks;
7. The patient is not required to have measurable systemic lesions; if there is, the lesions are required to be in at least one dimension (the largest diameter recorded by non-nodular lesions and the short axis of nodular lesions) ≥10mm by conventional techniques (CT, MRI) Can be accurately measured under the circumstances;
8. The subject himself voluntarily participated and signed an informed consent form.

Queue 2

1. Male or female,age at least 18 years ;
2. Histologically confirmed NSCLC patients (including patients who have relapsed after previous treatment or newly diagnosed);
3. Tumor cells found in cerebrospinal fluid or MRI showed clear meningeal enhancement and patients with dizziness/headache were included as selection criteria;
4. Patients who have not received other systemic treatment after being diagnosed with stage IV NSCLC, or patients who have received neoadjuvant therapy, adjuvant therapy, and concurrent radiotherapy and chemotherapy for more than 6 months;
5. The tumor tissue samples or blood are confirmed to be EGFR sensitive mutations (including exon 19 deletion or L858R) by ARMS;
6. The Eastern Cooperative Oncology Group (ECOG) physical status score is 0-2 and has not deteriorated in the previous 2 weeks, with a minimum expected survival of 12 weeks;
7. The patient is not required to have measurable systemic lesions; if there is, the lesions are required to be in at least one dimension (the largest diameter recorded by non-nodular lesions and the short axis of nodular lesions) ≥10mm by conventional techniques (CT, MRI) Can be accurately measured under the circumstances; The subjects themselves participated voluntarily and signed a written informed consent form.

Queue 3

1. Male or female,age at least 18 years ;
2. Histologically confirmed patients with stage IV NSCLC (including relapsed or newly diagnosed stage IV patients after previous treatment);
3. Patients with brain progression or brain lesions that have not resolved after the first/second generation EGFR-TKI treatment;
4. The patient must have at least one measurable brain lesion that has not been locally treated at the time of enrollment;
5. The tumor tissue samples or blood are confirmed to be EGFR sensitive mutations (including exon 19 deletion or L858R) by ARMS;
6. The Eastern Cooperative Oncology Group (ECOG) physical status score is 0-2 and has not deteriorated in the previous 2 weeks, with a minimum expected survival of 12 weeks;
7. The patient is not required to have measurable systemic lesions; if there is, the lesions are required to be in at least one dimension (the largest diameter recorded by non-nodular lesions and the short axis of nodular lesions) ≥10mm by conventional techniques (CT, MRI) Can be accurately measured under the circumstances;
8. The subject himself voluntarily participated and signed an informed consent form.

Exclusion Criteria:

1. the researchers believe that the risks faced by patients after entering the group are greater than those who benefit from them.
2. patients involved in any other clinical study.
3. patients with other malignant tumors.
4. A history of allergic reactions caused by compounds similar to almonertinib or its chemical composition.
5. pregnant or lactating women.
6. researchers should not participate in the study if they believe that patients cannot comply with the research procedures and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2023-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
iPFS | Up to approximately 3 years after the last patient is randomized
  Intracranial progression-free survival (iPFS)

SECONDARY OUTCOMES:
DCR | Up to approximately 3 years after the last patient is randomized
  Disease control rate (DCR)
PFS | Up to approximately 3 years after the last patient is randomized
  progression-free period (PFS)
OS | Up to approximately 3 years after the last patient is randomized
  overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Huijuan Wang, MD, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No